CLINICAL TRIAL: NCT00171847
Title: An Open Label, Randomized Comparison of Femara® 2.5mg Once Daily With or Without Weekly Herceptin® Until Disease Progression as First-line Treatment in Postmenopausal Women With Advanced Breast Cancer.
Brief Title: Study of the Efficacy and Safety of Letrozole Combined With Trastuzumab in Patients With Metastatic Breast Cancer
Acronym: eLEcTRA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Roche - Prof. Dr. Jens Huober et al. (Unknown)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345C2403
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2010-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; Metastatic; Trastuzumab; Letrozole
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Letrozole; Trastuzumab

ARMS (3):
- A - HER-2 +ve patients with Femara alone (Experimental)
  Interventions: Drug: Letrozole
- B - HER-2 +ve patients with Femara + Herceptin (Experimental)
  Interventions: Drug: Trastuzumab plus Letrozole
- C - HER-2 -ve patients with Femara alone (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Arms: A - HER-2 +ve patients with Femara alone
Drug: Trastuzumab plus Letrozole
  Arms: B - HER-2 +ve patients with Femara + Herceptin
Drug: Letrozole
  Arms: C - HER-2 -ve patients with Femara alone

SUMMARY:
Phase IV trial to investigate the effect of the combination of Letrozole with trastuzumab in metastatic breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Her-2 overexpression and ER and/or PgR positive
* Metastatic Breast Cancer

Exclusion Criteria:

* Previous treatment with trastuzumab
* Significant Liver or renal impairment
* Erbb2 negative and/or ER and PgR negative

Other protocol-defined inclusion / exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2003-03; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Time to progression as assessed by clinical palpation and radiologic imaging every 3 months | 3 months

SECONDARY OUTCOMES:
Objective response rate/Clinical Benefit rate | 3 months
Time to treatment failure | 3 months
Duration of response/clinical benefit during treatment | 3 months
Overall survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- Novartis Investigative Site, Tübingen, Germany